CLINICAL TRIAL: NCT03756285
Title: A Randomized, Double Blind, Placebo-controlled, Parallel Group, Multicentre, Phase 2a Study to Assess Target Engagement, Safety and Tolerability of AZD4831 in Patients With Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Safety and Tolerability Study of AZD4831 in Patients With Heart Failure.
Acronym: SATELLITE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A decision was made to stop the study early when AstraZeneca evaluated the available data and it was considered that completing the study would provide limited additional information and unlikely to change the study conclusions.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D6580C00003
Record Dates: First submitted 2018-11-19; First posted 2018-11-28 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Heart Failure
Keywords: Heart Failure with Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — AZD4831

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AZD4831 (Experimental): AZD4831 tablets taken orally for for 90 days.
  Interventions: Drug: AZD4831
- Placebo (Placebo Comparator): Placebo tablets taken orally for 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4831 — AZD4831 tablet taken orally for 90 days.
  Arms: AZD4831
Drug: Placebo — Placebo tablet taken orally for 90 days.
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel group, multicentre study in patients with Heart Failure with preserved Ejection Fraction (HFpEF). The study will be conducted at approximately 15 sites in 5 countries. Approximately 96 patients will be randomized to AZD4831 or placebo (treatment duration 90 days).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, parallel group, multicentre study in patients with Heart Failure with preserved Ejection Fraction (HFpEF) and mid-range Ejection Fraction (HRmrEF). The study will be conducted at approximately 15 sites in 5 countries (USA, Sweden, Denmark, Finland, Netherlands). Patients suitable for the study will be checked for eligibility, signing the informed consent and enrolled to the study at visit 1. The study will be divided into two parts, Part A and Part B. In part A 37 patients will be randomized at visit 2 in a 2:1 ratio to once daily dosing of AZD4831 or matching placebo for approximately 90 days. After approximately 30 days of treatment, an interim analysis will be done to analyse the safety, tolerability and target engagement. After the evaluation, the randomization to Part B may proceed. In Part B the approximate 59 remaining patients will be randomized and treated for approximately 90 days.

ELIGIBILITY:
Inclusion Criteria:

Informed consent

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this CSP
2. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses

   Age
3. Patient must be 45 to 85 years of age inclusive, at the time of signing the informed consent form

   Type of patient and disease characteristics
4. Signs and symptoms of HF in judgement of Investigator AND

   1. Stable NYHA II-IV and
   2. Ejection fraction (EF) ≥ 40 % and
   3. Elevated NT-proBNP or BNP in the last 1 year defined as:

      o Measured as out-patient: NT-proBNP ≥125 ng/L or BNP≥35 ng/L with sinus rhythm, NT-proBNP ≥750 ng/L or BNP ≥200 ng/L with atrial fibrillation (AF),

      or

      o Measured when hospitalized acutely: NT-proBNP ≥500 (ng/L) or BNP ≥125 ng/L with sinus rhythm, NT-proBNP ≥1250 (ng/L) or BNP ≥350 ng/L with AF
   4. And at least one of the following:

      * Hospitalization with HF as primary cause in last 12 months
      * Structural heart disease on echo according to ESC guidelines i.e. either enlarged Left atrial volume index (LAVI > 34 ml/m2) or increased LVM (LVM index > 95 g/m2 in women and > 115 g/m2 in men)
      * Pulmonary capillary wedge pressure (PCWP) at rest >15 mmHg or >25 mmHg at exercise
      * Spectral tissue Doppler echocardiography - E/e' ratio ≥13 at rest

   Weight
5. Body Mass Index (BMI) range 18-40kg/m2

   Sex
6. Male or female of nonchildbearing potential

   Reproduction
7. Female patients must be 1 year post-menopausal or surgically sterile
8. Male patients must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of AZD4831/matching placebo to prevent pregnancy in a partner. Male patients must not donate or bank sperm during this same time period

   Genetic sampling
9. For inclusion in this genetic research, patients must fulfil all of the inclusion criteria described above and provide informed consent for the genetic sampling and analysis

Exclusion Criteria:

Creatinine clearance by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) eGFR <30 ml/min/1.73m2 or dialysis

Life expectancy < 3 years due to other reasons than cardiovascular disease

Any ongoing skin disorder, history of or ongoing clinically significant allergy/hypersensitivity.

Current decompensated HF

Primary cardiomyopathy (e.g. constrictive, restrictive, infiltrative, toxic, hypertrophic, congenital or any primary cardiomyopathy) in judgment of investigator

Current hemodynamically significant valve disease in opinion of investigator

EF ever documented < 40%

Any current life-threatening dysrhythmia

Probable alternative primary reason for patient's symptoms in judgment of investigator, including but not limited to:

1. Isolated pulmonary arterial hypertension or right ventricular (RV) failure; in the absence of left-sided HF
2. Anaemia: Hb <100 mg/L (10g/dL)
3. Severe chronic obstructive pulmonary disease (COPD) or lung disease (chronic O2, nebulizer or oral steroid therapy)

Cardiac surgery, acute coronary syndrome (ACS), or non-elective percutaneous coronary intervention (PCI) < 3 months

Known or clinically judged significant macrovascular coronary artery disease (CAD) that has not been revascularized

Heart transplantation or left ventricular assist device ever

Patients with uncontrolled or clinically significant thyroid disease as judged by the investigator.

Alanine transaminase (ALT) or aspartate aminotransferase (AST) ≥2 x upper limit of normal (ULN). Resampling will not be allowed during the same screening period if detected abnormal values do not have reasonable explanation and are not expected to return to normal level within few days.

Known positive HIV, hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody, at screening

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (2):
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
- Denmark (4):
  - Research Site, Aarhus N
  - Research Site, Herlev
  - Research Site, Hvidovre
  - Research Site, Odense C
- Research Site, Turku, Finland
- Netherlands (3):
  - Research Site, Deventer
  - Research Site, Dordrecht
  - Research Site, Groningen
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Lam CSP, Lund LH, Shah SJ, Voors AA, Erlinge D, Saraste A, Pirazzi C, Grove EL, Barasa A, Schou M, Aziz A, Svedlund S, Wijngaarden JV, Lindstedt EL, Gustavsson A, Nelander K, Garkaviy P, Gan LM, Gabrielsen A. Myeloperoxidase Inhibition in Heart Failure With Preserved or Mildly Reduced Ejection Fraction: SATELLITE Trial Results. J Card Fail. 2024 Jan;30(1):104-110. doi: 10.1016/j.cardfail.2023.04.003. Epub 2023 Apr 16. PMID 37072105
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6580C00003&attachmentIdentifier=6f208598-cedf-467b-b3ef-41daf9951f1d&fileName=D6580C00003_CSP_redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6580C00003&attachmentIdentifier=2ff3c524-3bff-46d8-b76d-c14d8c93cefd&fileName=D6580C00003_SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZD4831 | Placebo
Started | 27 | 14
Completed | 24 | 9
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Study discontinued due to Other (Protocol deviation:subject meets exclusion criteria 20.) | 0 | 1
Not completed — Study discontinued due to Other (Dosing discontinued due to COVID-19) | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD4831 | Placebo | Total
Number analyzed (Participants) | 27 | 14 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (6.61) | 73.5 (6.99) | 74.3 (6.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 15 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 14 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 27 | 13 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Country [Count of Participants; unit: Participants]
  Denmark | 3 | 2 | 5
  Netherlands | 2 | 1 | 3
  USA | 0 | 1 | 1
  Finland | 5 | 3 | 8
  Sweden | 17 | 7 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MPO Specific Activity
Description: To compare the effect of AZD4831 to placebo on Target engagement, defined as ex vivo zymozan stimulated Myeloperoxidase (MPO) specific activity
Time Frame: Measurements on day 0, 10, 30 and 90. Change reported from day 0 to day 90.
Population: 20 of 27 patients in AZD4831 and 14 of 14 patients in placebo with evaluable measurements for analysis
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Groups:
- AZD4831: AZD4831 tablets taken orally for 90 days.
Arm/Group | AZD4831 | Placebo
Number analyzed (Participants) | 20 | 14
Ratio | 0.547 [0.379 to 0.790] | 2.177 [1.168 to 4.058]
Statistical Analysis 1: Comparison: AZD4831 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Covariates: atrial fibrillation status at randomization, baseline value, treatment, visit, and treatment*visit; Least Square Means Ratio = 0.25, 95% CI 2-sided [0.12 to 0.52]

2. Secondary Outcome: Change From Baseline in CFVR Measured in the Mid-distal Segment of the Left Anterior Descending (LAD) Coronary Artery Under Adenosine Infusion Measured by Transthoracic Doppler Echocardiography (TDE).
Description: To compare the effect of AZD4831 to placebo on coronary flow velocity reserve (CFVR) measured in the mid-distal segment of the left anterior descending (LAD) coronary artery under adenosine infusion measured by Transthoracic Doppler Echocardiography (TDE).
Time Frame: Measurement on day 0 and 90.
Population: 18 of 27 patients in AZD4831 and 5 of 14 patients in placebo with evaluable measurements for analysis
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | AZD4831 | Placebo
Number analyzed (Participants) | 18 | 5
Ratio | 0.975 [0.835 to 1.138] | 1.002 [0.747 to 1.344]
Statistical Analysis 1: Comparison: AZD4831 vs Placebo; Test type: Superiority; p = 0.568, ANCOVA; Covariates: atrial fibrillation status at randomization, baseline value, treatment; Least Square Means Ratio = 0.97, 95% CI 1-sided [lower limit 0.74]

3. Secondary Outcome: Change From Baseline in Walking Distance
Description: To compare the effect of AZD4831 to placebo on 6 minutes walking test (6MWT)
Time Frame: Measurement on day 0, 30 and 90. Change reported from day 0 to day 90.
Population: 23 of 27 patients in AZD4831 and 11 of 14 patients in placebo with evaluable measurements for analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: Meters
Arm/Group | AZD4831 | Placebo
Number analyzed (Participants) | 23 | 11
Meters | 47.4 [20.3 to 74.5] | 25.6 [-19.8 to 71.1]
Statistical Analysis 1: Comparison: AZD4831 vs Placebo; Test type: Superiority; p = 0.407, Mixed Models Analysis; Covariates: atrial fibrillation status at randomization, baseline value, treatment, visit, and treatment*visit; Mean Difference (Final Values) = 21.8, 95% CI 2-sided [-30.5 to 74.1]

ADVERSE EVENTS:
Time Frame: Adverse Events will be collected from the time of the first dose throughout the treatment period and including the follow-up period, up to 124 days. Serious Adverse Events will be recorded from the time of signing the informed consent form through follow-up period, up to 124 days.
Arm/Group | AZD4831 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/27 | 2/14
Other Adverse Events (participants affected / at risk) | 21/27 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD4831 (N=27) | Placebo (N=14)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD4831 (N=27) | Placebo (N=14)
Gingivitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Gout (Metabolism and nutrition disorders) | 2 | 0
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Blindness (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Infusion site oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Blood urea increased (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Troponin T increased (Investigations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Plicated tongue (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to premature study termination, the statistical assumptions for the study design according to the Clinical Study Protocol could not be fulfilled, therefore, no statistical conclusions can be made based on primary or secondary efficacy objectives. Statistical significance could not be evaluated for any efficacy objectives and the p-values presented are viewed as nominal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT03756285/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT03756285/SAP_001.pdf